CLINICAL TRIAL: NCT06473662
Title: A Phase 2b, Open-label Randomized Comparative Study to Evaluate the Safety and Efficacy of Oral Insulin Formulation in Type 2 Diabetes Mellitus Subjects Uncontrolled With Metformin Hydrochloride Treatment
Brief Title: Study to Evaluate the Safety and Efficacy of Oral Insulin Formulation in Type 2 Diabetes Mellitus Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roger New (Industry)
Responsible Party: Sponsor-Investigator, Roger New, Chief Scientific Officer, Diabetology Limited
Organization: Diabetology Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diabetology Ltd
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Treated With Insulin
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: A randomised twelve-week open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 75iu (Experimental): Capsule containing 75iu recombinant human insulin administered two times per day
  Interventions: Drug: Oral insulin
- 150iu (Experimental): Capsule containing 150iu recombinant human insulin administered two times per day
  Interventions: Drug: Oral insulin
- 300iu (Experimental): Capsule containing 300iu recombinant human insulin administered two times per day
  Interventions: Drug: Oral insulin

INTERVENTIONS:
Drug: Oral insulin — Capsule administered by mouth with a glass of water two times per day, once before breakfast and once before supper

SUMMARY:
The aim of the study was to compare the pharmacodynamic properties of different doses of regular human insulin administered in capsule form twice daily in a randomised twelve-week open-label trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 35 to 60 years (both inclusive)
2. Type 2 diabetes mellitus diagnosed < 2 years prior to enrolment
3. Glycated haemoglobin level ≥ 7% and ≤ 9.5%
4. On stable oral monotherapy with metformin hydrochloride (1000 mg to 2500 mg/day) and regular diet and exercise regimen at least 12 weeks prior to enrolment
5. Body mass index between 18 to 30 kg/m2
6. Ability to perform capillary blood glucose measurements
7. Willing to provide informed and written consent for the clinical trial
8. Able to comply with all requirements of clinical trial protocol

Exclusion Criteria:

1. Subject with history or evidence of hypersensitivity to insulin or metformin hydrochloride or its excipients
2. Suffering from type 1 diabetes mellitus
3. Received treatment with sulphonylureas or alpha-glucosidase inhibitors, Glucagonlike peptide-1 (GLP-1) receptor agonists or Sodium-glucose co-transporter 2 (SGLT2) inhibitors or meglitinides or pramlintide or thiazolidinediones within 3 months prior to enrolment
4. Previously treated with insulin within 3 months prior to enrolment
5. History of episodes of hypoglycaemia during 3 months prior to enrolment.
6. Reduced awareness of hypoglycaemia or inability to identify and tackle hypoglycaemic episodes
7. History of substantial weight loss defined as 5% decrease in body weight within the last 6 months
8. Medical history of unstable angina within 1 year prior to enrolment
9. History of tobacco or nicotine more than two packs/day within 3 months prior to enrolment
10. Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within 1 year prior to enrolment) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking).
11. History of gastrointestinal disorders which may potentially interfere with absorption of the investigational product
12. Treatment with systemic corticosteroids or with inhalational corticosteroids (Beclomethasone or budesonide) within the 3 months prior to enrolment
13. Likelihood of requiring treatment during the study period with prohibited medications mentioned (as defined in this clinical trial protocol)
14. Female subject who is pregnant, lactating or planning pregnancy during the trial
15. Female subject of childbearing age who is not willing to use adequate method of contraception during the study period
16. Life expectancy of less than 6 months from screening
17. Elective surgery or any other surgical procedure/s requiring general anaesthesia during the clinical trial
18. Has participated in another research trial within 12 weeks prior to screening
19. History of diabetic ketoacidosis requiring hospitalization within 6 months prior to enrolment, case of proliferative retinopathy or advanced neuropathy

    1. Subject having any of the following laboratory results at screening
    2. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2
    3. Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) >3 times of upper limit normal
20. Blood urea nitrogen (BUN) > 30 mg/dL
21. Subject who has a positive serology for hepatitis B virus (HBV) or hepatitis C (HCV) or human immunodeficiency virus (HIV) infections at screening
22. Subject who has undergone pancreatectomy or pancreas islet transplant or renal transplant
23. Subject receiving or has received any immunomodulation medications within 1 year prior to enrolment
24. Subject with history or evidence of diabetic complications (e.g. diabetic retinopathy, diabetic neuropathy, or diabetic nephropathy, etc.), cardiac disorders, or any other systemic complication due to diabetes, which in the opinion of the Investigator signifies subjects' ineligibility for the trial
25. Has any concurrent disease or medical/surgical condition, which required treatment of more than 3 months and which in the opinion of the Investigator does not allow participation of the subject in this study

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetology, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 204 patients were assessed for eligibility - 51 did not meet the inclusion criteria. Recruitment was conducted in hospital clinics and commenced one month before the start of study in October 2018
Pre-assignment Details: 153 patients were randomised to allocated treatment groups. A proportion of these patients (7) did not commence treatment, and full baseline characteristics were not collected for the whole group
Period: Overall Study
Arm/Group | 75iu | 150iu | 300iu
Started | 51 | 50 | 52
Completed | 33 | 29 | 38
Not Completed | 18 | 21 | 14
Not completed — Withdrawal by Subject | 1 | 6 | 5
Not completed — Uncontrolled hyperglycaemia | 1 | 2 | 2
Not completed — Starting HbA1c below 7% | 0 | 1 | 1
Not completed — No data from Central lab (protocol violation) | 14 | 9 | 4
Not completed — Did not take medication | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the number of patients who completed the study according to protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | 75iu | 150iu | 300iu | Total
Number analyzed (Participants) | 33 | 29 | 38 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 29 | 38 | 100
  >=65 years | 0 | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: years] | 48.8 (6.4) | 46.6 (6.3) | 49.7 (7.1) | 48.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 16 | 52
  Male | 13 | 13 | 22 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All patients in the population were of Indian origin, in accord with the location where the study was being caried out
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 33 | 29 | 38 | 100
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 33 | 29 | 38 | 100
HbA1c (%) [Mean (Standard Deviation); unit: %] | 8.27 (0.66) | 8.13 (0.65) | 7.93 (0.61) | 8.1 (0.65)
Body weight (kg) [Mean (Standard Deviation); unit: kg] | 63.9 (8.3) | 66.1 (8.8) | 66.9 (12.5) | 65.7 (10.2)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 25.6 (3.0) | 25.8 (2.7) | 25.7 (2.9) | 25.7 (2.8)
Fasting plasma glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 148.8 (53.0) | 148.2 (39.0) | 136.7 (47.8) | 144.0 (47.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in HbA1c Relative to Baseline at Start of Study
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of glycated haemoglobin
Arm/Group | 75iu | 150iu | 300iu
Number analyzed (Participants) | 33 | 29 | 38
% of glycated haemoglobin | -0.20 (1.06) | -0.53 (1.04) | -0.31 (1.04)
Statistical Analysis 1: Comparison: 150iu; Test type: Other; p = 0.0039, t-test, 2 sided; Mean Difference (Final Values) = -0.53

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in Fasting Plasma Glucose Relative to Baseline at Start of Study
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 75iu | 150iu | 300iu
Number analyzed (Participants) | 33 | 29 | 38
mg/dL | -14.8 (53.6) | -18.8 (39.8) | -2.7 (60.09)
Statistical Analysis 1: Comparison: 150iu; Test type: Other; p = 0.0166, t-test, 2 sided; Mean Difference (Final Values) = -18.8

3. Secondary Outcome: Change in Post-Prandial Glucose
Description: Change in Post-Prandial Glucose Relative to Baseline at Start of study
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 75iu | 150iu | 300iu
Number analyzed (Participants) | 33 | 29 | 38
mg/dL | -17.4 (83.74) | -21.0 (86.4) | -31.0 (97.7)

4. Secondary Outcome: Changes in Triglycerides
Description: Change in Triglycerides Relative to Baseline at Start of Study
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 75iu | 150iu | 300iu
Number analyzed (Participants) | 33 | 29 | 38
mg/dL | -7.06 (10.23) | -22.13 (11.02) | 20.56 (9.61)
Statistical Analysis 1: Comparison: 150iu; Test type: Other; p = 0.0474, ANCOVA; Mean Difference (Final Values) = -22.13

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 75iu | 150iu | 300iu
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29 | 0/38
Other Adverse Events (participants affected / at risk) | 0/33 | 0/29 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT06473662/Prot_SAP_000.pdf